CLINICAL TRIAL: NCT06189300
Title: The Effect of Telephone Education and Counseling to Individuals With Stoma on Stoma Compliance and Complications: Randomized Controlled Study
Brief Title: The Effect of Education and Counseling Given to People With Stoma by Telephone on Stoma Compliance and Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Seyma Yurtseven, Clinic Nurse, Cukurova University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 5077606250
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Stoma Colostomy
MeSH Terms: interventions — Educational Status; Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telephone Education (Experimental): Training and consultancy will be provided
  Interventions: Other: Education and counseling intervention
- Control (No Intervention): Standard care will be given

INTERVENTIONS:
Other: Education and counseling intervention — In addition to standard training, training and consultancy will be provided to individuals with stoma intermittently within a month.
  Arms: Telephone Education

SUMMARY:
The study will be conducted on individuals with stoma followed in the stoma therapy outpatient clinic of a university hospital. The effect size was found to be high, and the statistical power of the study was calculated as 2.955. Therefore, the power level was set at 0.80. The sample size for each group was calculated as 30 using the G*Power 3.1.9.7 program with an effect size of 0.8, 5% margin of error and 80% power %. Considering the possibility of data loss, the number of samples for each group was increased by 20% and it was planned to include 36 patients for each group. The Ostomy Adjustment Inventory and Pittman Ostomy Complication Severity Index will be completed. The scales will be collected for both groups on the first day, first month, and third month postoperatively. Patients were contacted five times postoperatively to provide education and counseling. SPSS will be used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Having undergone stoma surgery in a university hospital,
* No vision or hearing problems,
* Verbal communication is possible,
* Without diagnosed psychiatric problems.

Exclusion Criteria:

* Want to leave the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
The effect of education and counseling given to individuals with stoma on complications. | 1 and 3 mounth
  Pittman Ostomy Complication Severity Index will be used. This valid and reliable index was developed by Joyce Pittman in 2014 to evaluate the frequency and severity of complications developing in the early postoperative period during the follow-up period of individuals with a stoma. A higher total score indicates more serious ostomy complications. The lowest score that can be obtained from the scale is 0, while the highest score is 92.
The effect of education and counseling given to individuals with stoma on stoma compliance. | 1 and 3 mounth
  Ostomy Adjustment Inventory will be used. The lowest score that can be obtained from the scale is 0, while the highest score is 92.This valid and reliable scale was developed to determine the adaptation levels of individuals with stoma. A high score from the scale means that compliance is high.

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Adana, Turkey (Türkiye)